CLINICAL TRIAL: NCT03361189
Title: A Randomized Trial of Closed Loop Stimulation After Epicardial Pacemaker Implantation for Congenital Heart Disease
Brief Title: Specialized Pacing for Patients With Congenital Heart Disease
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: University of California, Los Angeles (Other)
Collaborators: Biotronik, Inc. (Industry)
Responsible Party: Principal Investigator, Jeremy P. Moore, MD, Associate Professor of Pediatrics, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 17-000932
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Results first posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-12

CONDITIONS: Congenital Heart Disease; Bradycardia Sinus
Keywords: Congenital heart disease; Pacemaker; Sinus node dysfunction
MeSH Terms: conditions — Heart Defects, Congenital; Sick Sinus Syndrome

STUDY DESIGN:
Intervention Model Description: Patient Enrollment: The treating physician will identify potential subjects with a previously implanted pacemaker and present a brief overview of the study. Informed consent will be obtained by the investigator after discussing the study, including the voluntary nature of participation and notification the subject can withdraw at any time. The investigator will give the subject and his/her legal guardian the opportunity to take the consent home to think about it more, with the option to call or meet with the investigator to ask additional questions. If the subject and/or his/her parent/legal guardian agree to participate, the investigator will ask them to sign a written, informed consent and assent.
  Randomization Procedure: This will be a single-blind placebo-controlled randomized crossover study with 2 treatments: CLS-on versus CLS-off (accelerometer only). Each enrolled patient will receive both treatments for 3 months. The order of treatments will be randomized 1:1.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CLS-On (Experimental): Subjects in this arm will be programmed to CLS-on to received closed loop stimulation-based pacing for 3 months, followed by a standard rate response for 3 months.
  Interventions: Device: Closed loop stimulation; Device: Standard rate response
- CLS-Off (Active Comparator): Subjects in this arm, will be placed in a standard rate response for 3 months, followed by CLS-on to received closed loop stimulation-based pacing for 3 months.
  Interventions: Device: Closed loop stimulation; Device: Standard rate response

INTERVENTIONS:
Device: Closed loop stimulation — Closed loop stimulation is a physiologic, rate-adaptive pacing algorithm.
Device: Standard rate response — Standard rate response is an algorithm to increase heartrate based on movement

SUMMARY:
The closed-loop stimulation (CLS) algorithm is a novel sensor-based technology that relies on the change in myocardial systolic impedance for modulation of the heart rate during physical and emotional stress.3 The pacing algorithm has been shown to be highly effective for a wide range of clinical scenarios. Despite the fact that congenital heart disease (CHD) patients are likely to derive significant benefit in terms of functional ability and aerobic capacity using this novel technology, the CLS system has not been adequately studied in this population. As many CHD patients also undergo epicardial placement of pacing systems at the time of concomitant cardiac surgery, CLS has been less often utilized in this population given almost no data in the setting of surgical electrode placement. The present study intends to examine the benefits of the CLS algorithm in the CHD population, employing the use of epicardial pacemaker systems in the study protocol.

DETAILED DESCRIPTION:
Sinus node dysfunction is highly prevalent among patients with congenital heart disease, manifesting as resting bradycardia or chronotropic incompetence. As children and adults with congenital heart disease are now expected to have increasing life-expectancy; with well over 1 million adult patients currently living in North America,1 issues such as mental health, acquired comorbidities and their impact on overall cardiovascular health have assumed increased scrutiny.

It is now understood that objective measures of aerobic capacity, such as peak VO2, peak VE/VCO2, and heart rate reserve predict all-cause mortality for adult patients with congenital heart disease. As the chronotropic response during exercise is a key determinant of aerobic capacity, improvement in sensor-based technology for heart rate support is expected to have a significant impact on functional capacity and longevity in this population. Some forms of congenital heart disease, such as single ventricle physiology after the Fontan population are especially likely to benefit, as cardiac output is determined almost exclusively by heart rate during exertion due to limited ability to augment cardiac stroke volume.2

It is also becoming increasingly clear that sedentary behaviors are highly relevant to overall cardiovascular health in the general adult population. Adult patients with congenital heart disease are at especially high risk for sedentary behavior as a result of 1) chronic restriction for physical activities based on ill-founded medical advice, 2) chronotropic incompetence resulting from prior surgical palliations and hemodynamic stressors, and 3) overestimation of physical activity.

5.0 Enrollment/Randomization

Patient Enrollment: The treating physician will identify potential subjects with a previously implanted pacemaker and present a brief overview of the study; if the subject is interested, the study will be described in detail. Informed consent will be obtained by the investigator after discussing the study, including the voluntary nature of participation and notification the subject can withdraw at any time. Ample time for questions and answers will be allowed. The investigator will give the subject and his/her legal guardian the opportunity to take the consent home to think about it more, with the option to call or meet with the investigator to ask additional questions. If the subject and/or his/her parent/legal guardian agree to participate, the investigator will ask them to sign a written, informed consent and assent. A copy of the assent and consent will be given to the subject and/or his/her parent/legal guardian.

Randomization Procedure: This will be a single-blind placebo-controlled randomized crossover study with 2 treatments: CLS-on versus CLS-off (accelerometer only). Each enrolled patient will receive both treatments for 3 months. The order of treatments will be randomized 1:1.

Randomization

There will be a 50:50 randomization, with half the subjects randomized to CLS-on then CLS-off, and half randomized to CLS-off then CLS-on.

Subjects previously receiving rate-responsive pacing with CLS that are randomly selected to CLS-on will continue with the identical programmed parameters. For subjects not previously receiving rate-responsive pacing with CLS that are randomly selected to CLS-on nominal programming will be utilized with a base rate of 60 beats per minute.

Subjects will then initiate treatment A (CLS-on or CLS-off) in a blinded fashion. At 3 months, subjects will undergo testing.

After 3 months of treatment A, subjects will be reprogrammed to treatment B. Tracking of physical activity with the device accelerometer will continue during this period. After 3 months of treatment B, repeat testing will be repeated.

Patients will be followed during both treatment phases per usual clinical routine. Patients who experience significant symptoms (extreme fatigue, debilitating palpitations, or other clinically relevant symptoms) will be evaluated by their treating physician. Subjects that have any adverse events during treatment A will discontinue treatment A and immediately crossover to treatment B. Subjects with events during treatment B will be removed from the study and unblinded. Further treatment will be determined by the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Congenital heart disease

  • Simple, moderate, or complex congenital heart disease
* Adolescent or adult age group (age >14 and <65 years)
* Significant sinus node dysfunction

  * Atrial pacing percentage >70%11
  * Intrinsic dysfunction resulting from congenital lesion or cardiac surgery
  * Secondary sinus node dysfunction due to antiarrhythmic drug therapy
* Existing, fully functional pacemaker or ICD with CLS capability
* Epicardial or transvenous route of pacemaker implantation

Exclusion Criteria:

* Unable to complete cardiopulmonary exercise testing (CPET)
* Contraindication to CPET
* Decreased mental capacity or known psychiatric disorder
* Congestive heart failure, NYHA cass IV
* Total atrial tachyarrhythmia burden >20%

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-05-09 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California at Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abi-Samra FM, Singh N, Rosin BL, Dwyer JV, Miller CD; CLEAR Study Investigators. Effect of rate-adaptive pacing on performance and physiological parameters during activities of daily living in the elderly: results from the CLEAR (Cylos Responds with Physiologic Rate Changes during Daily Activities) study. Europace. 2013 Jun;15(6):849-56. doi: 10.1093/europace/eus425. Epub 2013 Feb 17. PMID 23419655
- [Background] Bouchardy J, Therrien J, Pilote L, Ionescu-Ittu R, Martucci G, Bottega N, Marelli AJ. Atrial arrhythmias in adults with congenital heart disease. Circulation. 2009 Oct 27;120(17):1679-86. doi: 10.1161/CIRCULATIONAHA.109.866319. Epub 2009 Oct 12. PMID 19822808
- [Background] Chandiramani S, Cohorn LC, Chandiramani S. Heart rate changes during acute mental stress with closed loop stimulation: report on two single-blinded, pacemaker studies. Pacing Clin Electrophysiol. 2007 Aug;30(8):976-84. doi: 10.1111/j.1540-8159.2007.00795.x. PMID 17669080
- [Background] Coenen M, Malinowski K, Spitzer W, Schuchert A, Schmitz D, Anelli-Monti M, Maier SK, Estlinbaum W, Bauer A, Muehling H, Kalscheur F, Puerner K, Boergel J, Osswald S. Closed loop stimulation and accelerometer-based rate adaptation: results of the PROVIDE study. Europace. 2008 Mar;10(3):327-33. doi: 10.1093/europace/eun024. Epub 2008 Feb 13. PMID 18272507
- [Background] Di Pino A, Agati S, Bianca I. Efficacy of closed-loop stimulation with epicardial leads in an infant with congenital atrioventricular block. Europace. 2008 Mar;10(3):334-5. doi: 10.1093/europace/eum299. Epub 2008 Jan 20. PMID 18204100
- [Background] Hedman A, Nordlander R. Changes in QT and Q-aT intervals induced by mental and physical stress with fixed rate and atrial triggered ventricular inhibited cardiac pacing. Pacing Clin Electrophysiol. 1988 Oct;11(10):1426-31. doi: 10.1111/j.1540-8159.1988.tb04991.x. PMID 2462219
- [Background] Osswald S, Cron T, Gradel C, Hilti P, Lippert M, Strobel J, Schaldach M, Buser P, Pfisterer M. Closed-loop stimulation using intracardiac impedance as a sensor principle: correlation of right ventricular dP/dtmax and intracardiac impedance during dobutamine stress test. Pacing Clin Electrophysiol. 2000 Oct;23(10 Pt 1):1502-8. doi: 10.1046/j.1460-9592.2000.01502.x. PMID 11060870
- [Background] Quaglione R, Calcagnini G, Censi F, Piccirilli F, Iannucci L, Raveggi M, Biancalana G, Bartolini P. Autonomic function during closed loop stimulation and fixed rate pacing: heart rate variability analysis from 24-hour Holter recordings. Pacing Clin Electrophysiol. 2010 Mar;33(3):337-42. doi: 10.1111/j.1540-8159.2009.02615.x. Epub 2009 Nov 4. PMID 19889189
- [Background] Santini M, Ricci R, Pignalberi C, Biancalana G, Censi F, Calcagnini G, Bartolini P, Barbaro V. Effect of autonomic stressors on rate control in pacemakers using ventricular impedance signal. Pacing Clin Electrophysiol. 2004 Jan;27(1):24-32. doi: 10.1111/j.1540-8159.2004.00381.x. PMID 14720151
- [Background] Shachar GB, Fuhrman BP, Wang Y, Lucas RV Jr, Lock JE. Rest and exercise hemodynamics after the Fontan procedure. Circulation. 1982 Jun;65(6):1043-8. doi: 10.1161/01.cir.65.6.1043. PMID 7074766

RESULTS

PARTICIPANT FLOW:
Groups:
- CLS-On Followed by CLS-Off: Subjects in this arm will be programmed to CLS-on to received closed loop stimulation-based pacing for 3 months, followed by a standard rate response for 3 months.
  Closed loop stimulation: Closed loop stimulation is a physiologic, rate-adaptive pacing algorithm.
  Standard rate response: Standard rate response is an algorithm to increase heartrate based on movement
- CLS-Off Followed by CLS-On: Subjects in this arm, will be placed in a standard rate response for 3 months, followed by CLS-on to received closed loop stimulation-based pacing for 3 months.
  Closed loop stimulation: Closed loop stimulation is a physiologic, rate-adaptive pacing algorithm.
  Standard rate response: Standard rate response is an algorithm to increase heartrate based on movement
Period: Overall Study
Arm/Group | CLS-On Followed by CLS-Off | CLS-Off Followed by CLS-On
Started | 2 | 2
Completed Test Period 1 Completed | 1 | 1
Test Period 2 Begun | 1 | 1
Completed | 1 | 1
Not Completed | 1 | 1
Not completed — Received heart transplant | 1 | 0
Not completed — Pacemake replacement | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CLS-On Followed by CLS-Off | CLS-Off Followed by CLS-On | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Blunted or Unchanged Effect of Mental Stress on Heart Rate
Description: Heart rate in response to mental stress during each intervention; a math test was performed during autonomic testing
Time Frame: 3 months after the start of each intervention, a total of 6 months
Population: One participant completed autonomic testing
Measure: Count of Participants; unit: Participants
Groups:
- CLS-On: Subjects in this arm will be programmed to CLS-on to received closed loop stimulation-based pacing for 3 months Closed loop stimulation: Closed loop stimulation is a physiologic, rate-adaptive pacing algorithm.
- CLS-Off (Standard Rate Response): Subjects in this arm will be programmed to Standard rate response for 3 months. Standard rate response: Standard rate response is an algorithm to increase heartrate based on movement
Arm/Group | CLS-On | CLS-Off (Standard Rate Response)
Number analyzed (Participants) | 1 | 1
Participants
  Heart rate blunted | 1 | 0
  Heart rate unchanged | 0 | 1

2. Primary Outcome: Heart Rate Response During a 48-hour Assessment Period
Description: Average heart rate as measured by Holter monitor for 48 hours during each intervention
Time Frame: 3 months after the start of each intervention, a total of 6 months
Population: Participants with interpretable Holter monitor data under both interventions
Measure: Mean (Full Range); unit: beats per minute
Arm/Group | CLS-On | CLS-Off
Number analyzed (Participants) | 2 | 2
beats per minute | 74 [59 to 135] | 73 [40 to 144]

3. Secondary Outcome: Average Oxygen Consumption During Each Intervention
Description: Oxygen uptake as determined by cardiopulmonary gas exchange during a stress test under 4 conditions:
  Sitting/standing 60 seconds Kettlebell walking 110 seconds Stairs 176 seconds Sweeping 62 seconds
Time Frame: 3 months after the start of each intervention, a total of 6 months
Population: Only one participant completed stress tests, due to COVID restrictions, equipment and staffing issues
Measure: Number; unit: liters/minute
Arm/Group | CLS-On | CLS-Off
Number analyzed (Participants) | 1 | 1
liters/minute
  Sitting/Standing | 1.01 | 1.04
  Kettlebell walking | 1.02 | 1.10
  Stairs | 0.82 | 0.87
  Sweeping | 0.78 | 0.80

4. Secondary Outcome: Quality of Life as Assessed by SF-36
Description: Quality of life as assessed by SF-36 questionnaire following each period of intervetion. SF- 36 investigates the standard of quality of life through a general health assessment and not specific to a particular disease, age or treatment group. It is a 36-item questionnaire measuring 8 domains [physical functioning, role limitations due to physical health (role physical), bodily pain, general health, energy, social functioning, role limitations due to emotional health (role emotional), and emotional wellbeing]. Each domain score ranges from 0 (worst) to 100 (best), with higher scores reflecting better health-related functional status.
Time Frame: 3 months after the start of each intervention, a total of 6 months
Population: Two participants completed SF36 assessments
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | CLS-On | CLS-Off
Number analyzed (Participants) | 2 | 2
score on a scale
  Physical functioning | 95 [95 to 95] | 92.5 [90 to 95]
  Role physical | 100 [100 to 100] | 100 [100 to 100]
  Bodily pain | 90 [90 to 90] | 85 [80 to 90]
  General health | 67.5 [65 to 70] | 42.5 [35 to 50]
  Energy/vitality | 47.5 [35 to 60] | 47.5 [40 to 55]
  Social Function | 100 [100 to 100] | 100 [100 to 100]
  Role emotional | 100 [100 to 100] | 100 [100 to 100]
  Emotional wellbeing | 86 [84 to 88] | 84 [84 to 84]

ADVERSE EVENTS:
Time Frame: 3 months of each intervention
Groups:
- CLS-On: Participants received closed loop stimulation-based pacing (CLS-on) for 3 months.
  Closed loop stimulation: Closed loop stimulation is a physiologic, rate-adaptive pacing algorithm.
- CLS-Off: Participants received standard rate response (CLS-off) for 3 months.
  Standard rate response: Standard rate response is an algorithm to increase heartrate based on movement
Arm/Group | CLS-On | CLS-Off
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-01-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT03361189/Prot_SAP_002.pdf
  • Informed Consent Form (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT03361189/ICF_001.pdf